CLINICAL TRIAL: NCT00128570
Title: Cancer Prevention Mastery Model Internet Intervention
Brief Title: An Individualized Internet-Based Health Behavior Program or a Standard Internet-Based Health Behavior Program in Preventing Cancer and Improving Physical Activity and Nutrition in Participants Who Are Physically Inactive With a Higher Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000441158; VPISU-04-644; VPISU-03-588
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Early Intervention, Educational

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Other: educational intervention
Other: internet-based intervention
Other: preventative dietary intervention
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: An internet-based health behavior program that provides information about physical activity, fitness, and nutrition may help participants become healthier and reduce the risk of developing cancer.

PURPOSE: This randomized clinical trial is studying an individualized internet-based health behavior program to see how well it works compared to a standard internet-based health behavior program in preventing cancer and improving physical activity, fitness, and nutrition in participants who are physically inactive with a higher body mass index.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of an internet-based mastery-model health behavior educational intervention vs internet-based standard care health behavior educational intervention in improving physical activity and nutrition in sedentary participants with a higher body mass index.
* Compare the efficacy of these interventions in reducing cancer risk, in these participants.

OUTLINE: This is a randomized, controlled, multicenter study. Participants are stratified according to participating site, age (55 years and over vs under 55 years), gender, ethnic group, and aerobic capacity (≤ 6 metabolic equivalent tasks [METS] vs > 6 METS). Participants are randomized to 1 of 2 intervention arms.

* Arm I (mastery model health behavior educational intervention): Participants log on to the Guide to Health Project (GTH) website weekly and are provided access over a 24-month period to healthy lifestyle coaching modules and a completely individualized fitness program organized according to a mastery-model health behavior educational intervention. The mastery-model intervention comprises a 6-month behavioral initiation phase that includes an orientation and refinement of goals and expectations for each content area; a 6-month behavioral establishment phase comprising healthy lifestyle coaching modules focusing on physical activity and nutrition at least once a week; and a 6-month behavioral maintenance phase comprising a taper in the frequency of coaching sessions to once a month.
* Arm II (standard care health behavior educational intervention): Participants log on to the GTH website weekly and are provided access over a 24-month period to information regarding a healthy lifestyle focusing on physical activity and nutrition organized according to a standard care health behavior educational intervention.

In both arms, participants verify step-counts measured by a pedometer and complete the Block Food Frequency Questionnaire online at 10 and 18 months.

PROJECTED ACCRUAL: A total of 300 participants (150 per arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Sedentary participant

  * Not currently participating in a regular exercise program (i.e., < 30 minutes/day of moderate physical activity, 5 days a week)
* Body Mass Index 23-33.5
* Patiwnts that meet any of the following criteria are excluded:

  * High blood pressure (BP) (i.e., systolic BP ≥ 140 mm Hg OR diastolic BP ≥ 90 mm Hg) OR BP controlled with medications other than beta-blockers
  * Known high cholesterol (i.e., > 200 mg/dL)
  * Known low high-density lipoprotein level (i.e., < 40 mg/dL)
  * Use of antihyperlipidemic medications
  * Existing disease (i.e., heart disease, cancer, diabetes, and kidney or liver problems)

PATIENT CHARACTERISTICS:

Age

* 18 to 63

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No known liver disease

Renal

* No known kidney disease

Cardiovascular

* See Disease Characteristics
* No known cardiovascular disease
* Blood pressure ≤ 140/90 mm Hg

Pulmonary

* No known pulmonary disease

Other

* Not pregnant
* No known diabetes
* No known HIV positivity
* No cancer within the past 5 years
* No condition (e.g., orthopedic injuries or musculoskeletal disabilities) that would restrict physical activity or the ability to take a 1-mile walk test
* No other known life-threatening illness or condition
* Internet user

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior organ transplantation

Other

* No concurrent beta-blockers

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Winett, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

REFERENCES:
- [Result] Anderson-Bill ES, Winett RA, Wojcik JR. Social cognitive determinants of nutrition and physical activity among web-health users enrolling in an online intervention: the influence of social support, self-efficacy, outcome expectations, and self-regulation. J Med Internet Res. 2011 Mar 17;13(1):e28. doi: 10.2196/jmir.1551. PMID 21441100
- [Derived] Anderson-Bill ES, Winett RA, Wojcik JR, Winett SG. Web-based guide to health: relationship of theoretical variables to change in physical activity, nutrition and weight at 16-months. J Med Internet Res. 2011 Mar 4;13(1):e27. doi: 10.2196/jmir.1614. PMID 21447470